CLINICAL TRIAL: NCT02801903
Title: A Phase 1, Single-center, Open-label Pharmacokinetic, Safety and Tolerability Study of SB204 in Adolescents With Moderate to Severe Acne Vulgaris
Brief Title: Pharmacokinetics of Topical SB204 in Adolescents With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-AC103
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB204 4% (Experimental): Topically Once Daily (AM)
  Interventions: Drug: SB204 4%

INTERVENTIONS:
Drug: SB204 4% — Topically Once Daily (AM)
  Other Names: NVN1000

SUMMARY:
A Phase 1, Single-center, Open-label, Pharmacokinetic, Safety and Tolerability Study of SB204 in Adolescents with Moderate to Severe Acne Vulgaris

DETAILED DESCRIPTION:
This is a single-center, open-label study to be conducted in 18 otherwise healthy adolescents with moderate to severe acne vulgaris. Repeat blood samples will be obtained on Day 1 and Day 21 pre and post treatment to characterize systemic exposure to hMAP3 and nitrate. Subjects will receive a low-nitrate diet for 12 hours prior to and during the PK sampling period

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male and female adolescent subjects with moderate to severe acne vulgaris on a 5 point IGA scale
* At least 20 total inflammatory lesions (papules and pustules), and at least 20 total non-inflammatory lesions (open and closed comedones) on the face, chest, back, and shoulders
* Age 9-16 years, 11 months inclusive
* Subjects with methemoglobin level less than 3% at Screening and Baseline by pulse co-oximeter

Exclusion Criteria:

* Subjects with any other acne-like dermatological conditions such as severe, recalcitrant nodulocystic acne, acne conglobata, acne fulminans, acne secondary to medications or other medical conditions, perioral dermatitis, clinically significant rosacea, or gram-negative folliculitis;
* Any subject with skin disorders of an acute or chronic nature including psoriasis, eczema, tinea versicolor, etc.
* Subjects who reside in a dwelling that relies on well water for a primary drinking source
* Subjects with facial hair (beards, mustaches, etc.), tattoos or other facial markings that would interfere with assessments and study drug application
* Transgender subjects receiving hormone supplement (male to female or female to male)
* Subjects with a previous history of methemoglobinemia or taking medications known to be associated with methemoglobinemia
* Subjects with a known history of HIV, hepatitis, or other blood-borne pathogens
* Females who are pregnant, planning a pregnancy or breastfeeding
* Subjects previously treated with NVN1000 Gel / SB204

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of hMAP3 as measured by the maximum observed plasma concentration | Day 21
  Maximum plasma concentration of plasma hMAP3 on Day 21
AUC - area under the plasma concentration time curve for hMAP3 | Day 21
  AUC; area under the plasma concentration time curve from t=0 to the last measurable concentration for plasma hMAP3 on Day 21

SECONDARY OUTCOMES:
Pharmacokinetics as measured by maximum concentration of nitrate | Day 21
  Cmax: maximum plasma concentration of plasma nitrate on Day 21
Pharmacokinetics (AUC) - area under the plasma concentration time curve for hMAP3 | Day 21
  AUC; area under the plasma concentration time curve from t=0 to the last measurable concentration for plasma nitrate on Day 21
Safety profile (Reported adverse events) | Day 21/End of Treatment
  Reported adverse events
Tolerability (Scores on tolerability assessment) | Day 21/End of treatment
  Scores on tolerability assessment during treatment

CONTACTS AND LOCATIONS:
Overall Officials: M. Joyce Rico, MD, Study Director — Novan, Inc.
Locations (1):
- WCCT #1, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No